CLINICAL TRIAL: NCT00009243
Title: Evaluation, Pathogenesis, and Treatment of Patients With or at Risk for Cerebrovascular Disease (A Natural History/Disease Pathogenesis Protocol)
Brief Title: Natural History of Stroke: Cause and Development
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010007; 01-N-0007
Record Dates: First submitted 2001-01-24; First posted 2001-01-25 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-20

CONDITIONS: Brain Disease; Ischemic Attack, Transient; Cerebrovascular Accident; Cerebrovascular Disorder; Vascular Diseases
Keywords: Stroke; Natural History; MRI (Magnetic Resonance Imaging); Magnetic Resonance Imaging; Acute Stroke; TIA
MeSH Terms: conditions — Brain Diseases; Ischemic Attack, Transient; Stroke; Cerebrovascular Disorders; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with acute stroke symptoms

SUMMARY:
The purpose of this study is to learn more about stroke and obtain information that may serve as the basis for future investigations. It will 1) establish a registry of patients with cerebrovascular disease (stroke); 2) characterize the natural history of acute stroke and transient ischemic attacks (TIA)-an interruption of blood flow to the brain that causes stroke symptoms for a short period of time); and 3) evaluate the data to generate ideas for future studies.

Patients 18 years of age or older with suspected acute stroke or TIA may be eligible for this study. Subjects will be recruited from patients who present with stroke at the emergency department of Suburban Hospital in Bethesda, Maryland.

The study will gather data collected from diagnostic and laboratory tests the patient undergoes as part of standard medical care, including findings of medical and neurological examinations and other tests. In addition, studies will be done for research purposes only to gather data about stroke and TIA. These may include the following:

* Blood and urine tests not more than 2 tablespoons of blood will be drawn for various tests.
* Electrocardiogram (EKG) (heart tracing)-electrodes placed on the chest wall detect the heartbeat and heart rhythm.
* Computed tomography (CT) scan of the head-specialized X-rays are used to obtain images of the brain.
* Magnetic resonance imaging (MRI) of the brain-a strong magnetic field and radio waves are used to produce images that provide information about the brain tissue and blood vessels.
* Transcranial Doppler (TCD)-sound waves are used to image the arteries of the brain and neck.
* Echocardiogram-sound waves are used to image the heart and evaluate heart function.

Patients may be asked to return to Suburban Hospital for follow-up testing in 1, 3, and/or 12 months, when some of these tests may be repeated to assess changes over time

DETAILED DESCRIPTION:
Study Description:

This is a natural history/disease pathogenesis protocol for evaluation of patients with or at risk of acute stroke, transient ischemic attack (TIA), or other disturbances of cerebrovascular circulation. The purpose of this protocol is to generate natural history data to serve as the basis for future hypothesis-driven protocols as well as to contribute to the clinical and physiological understanding of cerebrovascular disease through the description of disease manifestation and the relationship among clinical, hematologic, and radiologic variables, as well as identifying potential subjects for future studies on stroke and other cerebrovascular diseases.

Objectives:

* To establish a registry of subjects with cerebrovascular disease including clinical, laboratory, and radiological variables associated with hemorrhagic and ischemic stroke, TIA, and other disturbances of cerebrovascular circulation.
* To characterize the natural history of acute stroke, TIA, and other disturbances of cerebrovascular circulation on these variables.
* To evaluate the relationship among these variables by exploratory analyses and to generate hypotheses for future testing.
* To identify potential subjects for research studies on stroke and other cerebrovascular diseases.

Endpoints:

A primary purpose of this observational protocol is to discover and study new imaging biomarkers that are i) relevant to the acute presentation and severity, ii) predictive of clinical outcome, and iii) are useful for stratifying the biological response as reflected in blood-biomarker and gene expression studies. As such, the primary outcome is the results from the imaging studies.

Primary Outcome Measures

Prevalence and type of abnormalities seen on neuroimaging as a function of time from acute insult such as:

* Imaging positive for acute ischemic cerebral vascular syndrome ( AICS positive )[1]
* Presence of a lesion on diffusion, perfusion, and mismatch between the two
* Evidence of a vascular occlusion on MR angiography
* Evidence of a thrombus or hemorrhage on T2* GRE imaging
* Blood-brain barrier disruption as evidence by HARM [2]
* The evolution of these markers with time and treatment

Secondary Outcome Measures

* Stroke severity as measured by NIHSS as a function of time since index event.
* Clinical outcome measured using modified Rankin Scale and Barthel Index
* Gene expression profiles and biomarker levels obtained from blood samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Aged >=18
2. Presented to participating study site (ED, ICU, or inpatient unit) with or at risk of acute stroke, TIA, or other disturbances of cerebrovascular circulation

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Subjects with contraindication to MRI scanning will be excluded from any testing which involves the use of MRI. The contraindications include subjects with the following devices or conditions:

   * Central nervous system aneurysm clips
   * Implanted neural stimulator
   * Implanted cardiac pacemaker or defibrillator
   * Cochlear implant
   * Ocular foreign body (e.g. metal shavings)
   * Insulin pump
   * Metal shrapnel or bullet
   * Any implanted device that is incompatible with MRI

   Subjects with a condition precluding entry in the scanner (e.g. morbid obesity, Claustrophobia, etc.) will not be included in the MRI portion of this study.
2. Pregnancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from the collaborative stroke programs between NINDS and affiliated hospitals (Suburban Hospital and MedStar Washington Hospital Center) and will be followed for the duration of their hospitalization. Select subjects will then be seen for follow up for up to one year.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2001-01-26 (Actual)

PRIMARY OUTCOMES:
Prevalence and type of abnormalities seen on neuroimaging as a function of time from acute insult | Post-acute, 24 hours, 5 days/discharge, 30 days
  Neuroimaging abnormalities, such as:-Imaging positive for acute ischemic cerebral vascular syndrome ( AICS positive )-Presence of a lesion on diffusion, perfusion, and mismatch between the two-Evidence of a vascular occlusion on MR angiography-Evidence of a thrombus or hemorrhage on T2* GRE imaging-Blood-brain barrier disruption as evidence by "HARM"-The evolution of these markers with time and treatment

SECONDARY OUTCOMES:
Stroke severity as measured by NIHSS as a function of time since index event | Post-acute, 24 hours, 5 days/discharge, 30 days, 3 months, 6 months, 12 months
Clinical outcome measured using modified Rankin Scale and Barthel Index | 5 days/discharge, 30 days, 3 months, 6 months, 12 months
Gene expression profiles and biomarker levels obtained from blood samples | Post-acute, 24 hours, 5 days/discharge, 30 days, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence L Latour, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (3):
- United States (3):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Suburban Hospital - Johns Hopkins Medicine, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie the results reported in the publication, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years after article publication.
Access Criteria: IPD will be shared with researchers who provide a methodologically sound proposal . Proposals should be sent to the corresponding author of the publication.

REFERENCES:
- [Derived] Lomahan CA, Luby M, Kalarakis G, Hsia AW, Lynch JK, Nathani KP, Somani S, Thomas LC, Arnberg-Sandor F, Latour LL. Hyperemia detection on arterial spin labeling is associated with final infarct volume in stroke post-endovascular therapy. J Stroke Cerebrovasc Dis. 2025 Aug;34(8):108358. doi: 10.1016/j.jstrokecerebrovasdis.2025.108358. Epub 2025 May 26. PMID 40436255
- [Derived] Cho YE, Lee H, Bae HR, Kim H, Yun S, Vorn R, Cashion A, Rucker MJ, Afzal M, Latour L, Gill J. Circulating immune cell landscape in patients who had mild ischaemic stroke. Stroke Vasc Neurol. 2022 Aug;7(4):319-327. doi: 10.1136/svn-2021-001224. Epub 2022 Mar 9. PMID 35264400
- [Derived] Luby M, Hsia AW, Nadareishvili Z, Cullison K, Pednekar N, Adil MM, Latour LL. Frequency of Blood-Brain Barrier Disruption Post-Endovascular Therapy and Multiple Thrombectomy Passes in Acute Ischemic Stroke Patients. Stroke. 2019 Aug;50(8):2241-2244. doi: 10.1161/STROKEAHA.119.025914. Epub 2019 Jun 26. PMID 31238832
- [Derived] Hsia AW, Luby M, Cullison K, Burton S, Armonda R, Liu AH, Leigh R, Nadareishvili Z, Benson RT, Lynch JK, Latour LL. Rapid Apparent Diffusion Coefficient Evolution After Early Revascularization. Stroke. 2019 Aug;50(8):2086-2092. doi: 10.1161/STROKEAHA.119.025784. Epub 2019 Jun 26. PMID 31238830
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-N-0007.html